CLINICAL TRIAL: NCT04039841
Title: Pilot Study to Predict Falls with Motor Imagery
Brief Title: Is It Possible to Predict Falls with Motor Imagery
Acronym: FallMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion was stopped prematurely on 18/01/2024, following a delay in inclusion that could not be made up within the regulatory timeframe. The final follow-ups were carried out in accordance with the protocol.
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CHD 032-18
Record Dates: First submitted 2019-07-22; First posted 2019-07-31 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Fall Patients

STUDY DESIGN:
Intervention Model Description: Non-interventional Monocentric Prospective Non-intervention Research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Motor imagery evaluation (Other): cohort study
  Interventions: Diagnostic Test: Motor Imagery Test

INTERVENTIONS:
Diagnostic Test: Motor Imagery Test — Imagined Timed Up and Go (iTUG) is the imagined version of the actual Timed Up and Go (rTUG) described above). It is possible to calculate the absolute value of the difference between the time of execution of the TUG imagined and actually executed. This difference is called isochrony index. The alteration of this isochrony index is correlated with the decrease in walking speed during the double task. This test is performed during the osteoporosis screening consultation.
  For patients who agree to participate in the FallMI study, the name and contact information of the attending physician will be collected during the same consultation.
  Standardised email will be sent to the attending physicians to collect the presence of falls and its consequences. They will be classified as fatal, severe, moderate and inconsequential.

SUMMARY:
At Departmental Hospital Centre, a primary and secondary screening program for osteoporosis was set up in 2014 in the medical services (excluding oncology), gynaecology, outpatient surgery and orthopaedics. Patients who consulted outpatients in the emergency room were not taken into account due to the 24-hour opening hours. The objective of this program was to identify all patients at risk of osteoporosis; i. e. not only patients with a recent or previous fracture history, but also patients with osteoporosis risk factors without a history of fracture to date. This is in order to propose a prevention strategy to referring physicians and thus reduce the risk of fractures. The handover of the Timed Up and Go designed and physically carried out was added in July 2017 to the management of patients as part of this screening.

During this screening, patients are asked to perform 2 realized Timed Up and Go (rTUG), followed by 2 imagined Timed Up and Go (iTUG).

The interest in preventing falls in osteoporotic patients leads investigators to propose this evaluation as part of this "osteoporosis" screening. The investigators will offer patients benefiting from osteoporosis screening as part of the process already in place at Departmental Hospital Centre to participate in the FallMi study. If agreement is reached, the patient's treating physician will be contacted to collect data on the occurrence of falls in these patients. After a request by mail, an email will be sent to the attending physicians of each patient at 6 months, then one year after the completion of the TUG. This email will ask physicians about the presence of a fall that has occurred since the TUGs were performed, as well as the severity of this possible fall.

Investigators objective is to evaluate rTUG and iTUG as predictive factors of a fall with moderate to fatal consequences.

Investigators hypothesize that a lower isochrony between rTUG and iTUG is predictive of a risk of falling.

DETAILED DESCRIPTION:
Fall of the elderly is a major public health problem, especially in people with fragile bones. Various tools are available to identify high-risk subjects. Timed Up and Go (TUG) is a clinical test used as a predictive test of fall. However, its real usefulness remains uncertain. The degradation of TUG appears to be validated after the fall, but discussed as a prediction of a future fall.

On the other hand, human movement is separable into 2 phases, a programming phase (anticipation) and an execution phase. Movement programming can be reliably assessed through a simple test that evaluates the concordance between the duration of an imagined practice and a physical practice . Adapted to Timed Up and Go (= |realizedTUG -imaginedTUG|), the degradation of this Isochronic Index clinically marks a structural and functional degradation of cognitive abilities . In addition, the decrease in isochrony is correlated with the decrease in walking speed during the double task. This loss of isochrony could thus indicate a risk of falling due to poor anticipation of real motor skills.

At Departmental Hospital Centre, a primary and secondary screening program for osteoporosis was set up in 2014 in the medical services (excluding oncology), gynaecology, outpatient surgery and orthopaedics. Patients who consulted outpatients in the emergency room were not taken into account due to the 24-hour opening hours. The objective of this program was to identify all patients at risk of osteoporosis; i. e. not only patients with a recent or previous fracture history, but also patients with osteoporosis risk factors without a history of fracture to date. This is in order to propose a prevention strategy to referring physicians and thus reduce the risk of fractures. The handover of the Timed Up and Go designed and physically carried out was added in July 2017 to the management of patients as part of this screening.

During this screening, patients are asked to perform 2 realized Timed Up and Go (rTUG), followed by 2 imagined Timed Up and Go (iTUG).

The interest in preventing falls in osteoporotic patients leads us to propose this evaluation as part of this "osteoporosis" screening. This study wills offer patients benefiting from osteoporosis screening as part of the process already in place at CHD to participate in the FallMi study. If agreement is reached, the patient's treating physician will be contacted to collect data on the occurrence of falls in these patients. After a request by mail, an email will be sent to the attending physicians of each patient at 6 months, then one year after the completion of the TUG. This email will ask the doctors about the presence of a fall that has occurred since the TUGs were performed, as well as the severity of this possible fall.

Investigators objective is to evaluate rTUG and iTUG as predictive factors of a fall with moderate to fatal consequences.

Investigators hypothesize that a lower isochrony between rTUG and iTUG is predictive of a risk of falling.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been screened for osteoporosis at CHD (aged 50 to 85 years)
* Proven presence of osteoporotic risk (positive response to screening tests),
* No lower limb fractures making walking impossible,
* Realization of iTUG and rTUG.
* No objection to the collection and analysis of personal data collected,
* Patient can be followed during the study period (12 months),
* Patient followed by a treating physician and having given his or her consent for him or her to be contacted as part of the study.

Exclusion Criteria:

* Insane patient
* Deaf patient
* Complete blind patient
* Patient unable to express himself
* Patient at the end of life
* Patient already treated for osteoporosis or recent DXA less than 3 years old at the time of screening
* Patient who has not been screened for osteoporosis at the CHD
* Presence of equipment (e.g. infusion) making it impossible to walk or rendering the reliability of TUGs obsolete,

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
existence of an isochronic deficit between the imagined Timed Up and Go and the Timed Up and Go correlated with presence of a fall | 6 month
  - Isochronic index =| rTUG-iTUG | (Absolute value of the difference between the execution time of the rTUG and the iTUG)

SECONDARY OUTCOMES:
Evaluate the factors that predict a fall | 12 month
  - Isochronic index =| rTUG-iTUG | (Absolute value of the difference between the execution time of the rTUG and the iTUG)
Assess the factors that predict a first fall | 6 and 12 month
  - Isochronic index =| rTUG-iTUG | (Absolute value of the difference between the execution time of the rTUG and the iTUG)
Assess whether factors are predictive of the severity of a fall | 6 and 12 month
  - Isochronic index =| rTUG-iTUG | (Absolute value of the difference between the execution time of the rTUG and the iTUG)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rulleau, PT PhD, Principal Investigator — CHD-Vendee
Locations (1):
- Centre Hospitalier Departemental, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No